CLINICAL TRIAL: NCT06751771
Title: Effects of Comprehensive Correcting Exercise Program and Mckenzie Exercises in Patients With Sternosymphyseal Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0109
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Sterno Sympheseal Syndrome
Keywords: Corrective exercises; McKenzie exercises; Thoracic kyphosis; Range of Motion; Functional Disability

STUDY DESIGN:
Intervention Model Description: COMPARATIVE EFFECTS OF COMPREHENSIVE CORRECTING EXERCISE PROGRAM AND MCKENZIE EXERCISES PROTOCOL ON PAIN, CRANIOVERTEBRAL ANGLE, THORACIC KYPHOSIS ANGLE, RANGE OF MOTION AND FUNCTIONAL DISABILITY IN PATIENTS WITH STERNOSYMPHYSEAL SYNDROME
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comprehensive correcting exercise program (Experimental): Group A will be treated with comprehensive correcting exercise program (three times a week for 6 weeks) into 3 phases with different intensity and frequency
  Interventions: Other: comprehensive correcting exercise program
- McKenzie's method of exercises (Experimental): Group B will receive the McKenzie's method of exercises that include Deep neck flexor (chin tucks), Shoulders shrug McKenzie exercise for neck, Repeated shoulder flexion/Extension, Neck flexion McKenzie exercises
  Interventions: Other: McKenzie's method of exercises

INTERVENTIONS:
Other: comprehensive correcting exercise program — Group A will be treated with comprehensive correcting exercise program (three times a week for 6 weeks) into 3 phases with different intensity and frequency
  Arms: comprehensive correcting exercise program
Other: McKenzie's method of exercises — Group B will receive the McKenzie's method of exercises that include Deep neck flexor (chin tucks), Shoulders shrug McKenzie exercise for neck, Repeated shoulder flexion/Extension, Neck flexion McKenzie exercises
  Arms: McKenzie's method of exercises

SUMMARY:
A Randomized Clinical Trial will be conducted at Horizon Hospital Physiotherapy Department and Riphah Clinic Lahore through consecutive sampling technique on 36 patients which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with comprehensive correcting exercise program (three times a week for 6 weeks) into 3 phases with different intensity and frequency. Group B will receive the McKenzie's method of exercises that include Deep neck flexor (chin tucks), Shoulders shrug McKenzie exercise for neck, Repeated shoulder flexion/Extension, Neck flexion McKenzie exercises. Outcome measure will be conducted through pain and functional disability Index through questionnaire and craniovertebral angle through PhysioMaster/APECS, Thoracic kyphosis through Inclinometer and Range of motion via goniometer.

DETAILED DESCRIPTION:
Sternosymphyseal syndrome is a postural syndrome involves excessive lumbar and thoracic kyphosis, a forward drawn head, and hyper-lordosis of the cervicocranial junction. This posture is associated with increased muscular tension and faulty respiration habits. When the slumped posture is assumed for sustained periods of time, increased load is placed on the intervertebral disc. With the sternum approximating the pubic symphysis, diaphragmatic inhibition results in over-activation of scalene and upper trapezius musculature during respiration. This muscle tension is reversible by merely having the patient sit up straight. (Brugger's relief position).

A Randomized Clinical Trial will be conducted at Horizon Hospital Physiotherapy Department and Riphah Clinic Lahore through consecutive sampling technique on 36 patients which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with comprehensive correcting exercise program (three times a week for 6 weeks) into 3 phases with different intensity and frequency. Group B will receive the McKenzie's method of exercises that include Deep neck flexor (chin tucks), Shoulders shrug McKenzie exercise for neck, Repeated shoulder flexion/Extension, Neck flexion McKenzie exercises. Outcome measure will be conducted through pain and functional disability Index through questionnaire and craniovertebral angle through PhysioMaster/APECS, Thoracic kyphosis through Inclinometer and Range of motion via goniometer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-28
* Both gender male and female
* Participants who have any distance from xiphoid process to pubic symphysis less than 18cm (11 inches)
* Participants with forward head (≥ 44°), round shoulder (≥ 49°) or excessive thoracic kyphosis (≥ 42°) will be measured by photography and flexicurve. Patient agree to sign written consent

Exclusion Criteria:

* Subjects younger than 18 years of age, cardiac, respiratory, kidney, circulatory problems, systemic disease, diabetes
* Any trauma or localized infection in neck region
* Pregnancy or suspicion of pregnancy for female subjects.
* A history of fractures, treatment or surgery to the lumbar, thoracic, cervical spine and upper limbs
* Thoracic outlet syndrome.
* Any shoulder pathology causing limitation of movement.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Inclinometer | 6 WEEK
  The thoracic kyphosis will be measured by using an inclinometer. The feet of inclinometer will be placed on the spinal vertebrae which will be palpated first
Numeric pain rate scale (NPRS) | 6th week
  Patient level of pain will be assessed using this 11-point NPRS scale (0-no pain, 10-most intense pain) is the most commonly used version which has good test-retest reliability (r=. 79-. 96) This scale ranges from 0 to 10

SECONDARY OUTCOMES:
Neck Disability Index | 6 WEEK
  This questionnaire will be used to assess disability. It comprises of 10 items; 7 related to daily living activities, 2 related to pain and 1 related to concentration. Each item is scored from 0 to 5. Total score is expressed as a percentage, with higher scores related to greater disability (24). The 10 items, with 6 possible answers in each are scored 0 (no activity limitations) to 5 (major activity limitations) and summed up to yield a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University
Locations (1):
- Physiotherapy department of Horizon Hospital and Riphah International clinic Lahore., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morris CE, Greenman PE, Bullock MI, Basmajian JV, Kobesova A. Vladimir Janda, MD, DSc: tribute to a master of rehabilitation. Spine (Phila Pa 1976). 2006 Apr 20;31(9):1060-4. doi: 10.1097/01.brs.0000214879.93102.4e. PMID 16641785
- [Background] Page P. Shoulder muscle imbalance and subacromial impingement syndrome in overhead athletes. Int J Sports Phys Ther. 2011 Mar;6(1):51-8. PMID 21655457
- [Background] Czaprowski D, Stolinski L, Tyrakowski M, Kozinoga M, Kotwicki T. Non-structural misalignments of body posture in the sagittal plane. Scoliosis Spinal Disord. 2018 Mar 5;13:6. doi: 10.1186/s13013-018-0151-5. eCollection 2018. PMID 29516039